CLINICAL TRIAL: NCT00784771
Title: Hypnotherapeutic Olfactory Conditioning for Chronic Combat-Related Posttraumatic Stress Disorder
Brief Title: Hypnotherapeutic Olfactory Conditioning for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzog Hospital (Other)
Responsible Party: Dr. Pesach Lichtenberg, Herzog Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lichtenberg4 CTIL
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Hypnotherapy; Hypnosis; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Hypnotherapeutic Olfactory Conditioning (HOC)

SUMMARY:
Chronic combat-related posttraumatic stress disorder can be difficult to treat. The investigators believe that hypnosis, with a stress on the sensation of scent which often plays a role in the traumatic memories, can offer help for victims of this disorder who continue to suffer after receiving other treatments.

DETAILED DESCRIPTION:
Our study examines the effect of hypnosis upon 36 individuals who suffer from posttraumatic stress disorder incurred in battles or training. The hypnotherapy stresses elements of odor, both in conditioning the subject to relate certain pleasant odors with security and calm, and in gradually reexposing the patient to the olfactory aspects of the traumatic memories. All subjects are taken form the Israel Defense Forces Mental Health Clinic, treated with 6 one-and-a-half-hour hypnotherapy sessions, and evaluated at baseline, end of treatment, after 6 months, and after 12 months, on a battery of clinical scales.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of chronic combat-related PTSD according to DSM-IV criteria (APA, 1994), as determined by semi-structured psychiatric interview conducted by a psychiatrist with over ten years of experience treating PTSD
2. Flashbacks and/or panic attacks with olfactory components
3. Prior attempt at treatment with unsatisfactory results
4. Competence and agreement to sign an informed consent.

Exclusion Criteria:

1. Evidence of psychosis
2. Severe traumatic brain injury
3. Post-concussion syndrome
4. Uncontrolled substance abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Impact of Event Scale | Baseline, 6 weeks, 6 months, one year

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline, 6 weeks, 6 months, one year
Dissociative Experience Scale | Baseline, 6 weeks, 6 months, one year

CONTACTS AND LOCATIONS:
Locations (1):
- Combat Stress Reaction Unit, Medical Corps, Mental Health Department, Israel Defense Forces, Tel Litwinsky, Ramat Gan, Israel